CLINICAL TRIAL: NCT07399964
Title: Effects of Cognitive Behavioural Therapy for Insomnia (CBT-I) on Impulsivity and Risk Taking in Youths With Insomnia: A Randomised Controlled Trial
Brief Title: Effects of CBT-I on Impulsivity and Risk Taking in Youths With Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); King's College London (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA230518
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Insomnia; Impulsivity; Risk-Taking
Keywords: Insomnia; Youth; Impulsivity; Inhibitory Control
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Impulsive Behavior; Risk-Taking | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental): N = 62
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia
- Health-related Psychoeducation control (Active Comparator): N = 62
  Interventions: Other: Health-related Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia — CBT-I consists of 6 weekly group sessions (90-min, 5-8 adolescents in each group) delivered in the afternoon/evening after school within a 10-week window. The intervention is structured and based on the well-established CBT elements for treating insomnia. The treatment components aim to address the behavioural, cognitive, and physiological factors perpetuating insomnia whilst considering the sleep and circadian features in adolescents and developmental context with the following key elements: psychoeducation about sleep, circadian rhythm and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Arms: CBT-I
Other: Health-related Psychoeducation — The active control group will receive group-based health-related psychoeducation, a format that has been adopted in the previous research, in order to provide the credibility of the intervention to the participants, and to control for the potential effects of attention and nonspecific components, e.g., receiving health-related information, expectations of benefit. It will also consist of 6 weekly sessions which contain education on general well-being, diet, and exercise/activity.
  Arms: Health-related Psychoeducation control

SUMMARY:
Insomnia is prevalent in adolescents. Impulsive behaviours and excessive risk-taking have been linked to the manifestation of psychopathology in youths. Previous research based on behavioural and neurophysiological measures has found that individuals with insomnia demonstrated impaired inhibitory control, which is associated with detrimental outcomes such as substance abuse and self-harm.

Existing evidence has shown some positive effects of cognitive behavioural therapy for insomnia (CBT-I) on insomnia symptoms and daytime functioning in youths. Given the link between insomnia and impulsivity reported in previous research, and sleep as a highly modifiable factor, we are conducting this randomised controlled trial to examine the impact of CBT-I in improving impulsivity and risk-taking in youth with insomnia.

DETAILED DESCRIPTION:
A randomised, assessor-blind, parallel-group controlled trial will be conducted on youths with insomnia. The study aims to test the effects of CBT-I on impulsivity in adolescents, as assessed through both self-report and objective measures when compared with the psychoeducation control. Eligible participants will be randomised to either group-based CBT-I or psychoeducation control condition. Randomisation will be carried out using an automated online system. Assessments will be conducted at pre-treatment (week 0) and post-treatment (week 7/one-week after the last group session), as well as post-treatment 6 months in order to examine the maintenance effects following the CBT-I intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chinese aged 12-24 years old
* Written informed consent of participation in the study is given by the participant and his/her parent or guardian (for those aged under 18)
* Willing to comply with the study protocol
* Meeting the DSM-V diagnostic criteria of insomnia disorder and with a score on Insomnia Severity Index (ISI) >= 9 (suggested cut-off for adolescents)

Exclusion Criteria:

* A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities
* Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema, gastro-oesophageal reflux disease)
* Having a clinically diagnosed sleep disorder (other than insomnia disorder) that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome, as ascertained by the Structured Interview for Sleep Patterns and Disorders (DISP), a validated structured diagnostic interview to assess major sleep disorders according to the International Classification of Sleep Disorder (ICSD) criteria
* Concurrent, regular use of medications(s) known to affect sleep continuity and quality including both western medications (e.g. hypnotics, steroids) and over-the-counter OTC medications (e.g. melatonin, Traditional Chinese Medicine, TCM)
* In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt)
* Currently receiving any psychological treatment for insomnia
* With hearing or speech deficit
* Night shift worker

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Impulsivity | Baseline, one week after the intervention and 6-month after the intervention
  Change in the degree of impulsivity is the degree will be measured by UPPS-P Impulsive Behavior Scale.

SECONDARY OUTCOMES:
Change in Insomnia Symptoms | Baseline, one week after the intervention and 6-month after the intervention
  Insomnia symptoms are measured by the Insomnia Severity Index (ISI). ISI is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.
Change of Sleep Diary Measure - Time in Bed (TIB) | Baseline, one week after the intervention and 6-month after the intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours.
Change of Sleep Diary Measure - Total Sleep Time (TST) | Baseline, one week after the intervention and 6-month after the intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours.
Change of Sleep Diary Measure - Sleep Onset Latency (SOL) | Baseline, one week after the intervention and 6-month after the intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins.
Change of Sleep Diary Measure - Sleep Efficiency (SE) | Baseline, one week after the intervention and 6-month after the intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %.
Change of Actigraphy- based Measure | Baseline, one week after the intervention and 6-month after the intervention
  Sleep-wake pattern will be objectively measured by 7-day wrist actigraphy (Actiwatch Spectrum, Philips Respironics). Sleep parameter estimated by actigraphy will include time in bed, total sleep time, sleep onset latency (SOL), wake after sleep onset (WASO), and sleep efficiency.
Change of Objective Cognitive Performance (Cued Go/NoGo) | Baseline, one week after the intervention and 6-month after the intervention
  The Cued Go/NoGo task is a spatial-cueing task with equal probability of Go and NoGo stimuli. In the beginning of each trial, a left or right pointing arrow is presented for 200ms as a cue, instructing the participants to attend to the cued location and ignore the other. Following interval varying from 1000-1200ms from cue offset, a target is presented for 200ms. Participants should respond to the plus sign '+' (Go) at the cued location (Attend-Go), whilst inhibit from responding to the letter 'x' (NoGo) at the cued location (Attend-NoGo). For any target appearing at the ignored location, participants should not respond to either the Go target (Ignore- Go) or the NoGo target (Ignore-NoGo). The percentage of errors in all the trials (total error), the percentage of errors in Attend-NoGo trials (commission errors, indicating inhibition error), and the reaction time in Attend-Go trials with accurate responses (reaction time).
Change of Objective Cognitive Performance (Balloon Analogue Risk Task) | Baseline, one week after the intervention and 6-month after the intervention
  In this task, participants are instructed to fill the balloon with air by selecting number of "pumps" on the dial. Once the number of pumps was selected, the balloon would automatically expand until the target pump number was reached or the balloon popped. Either a green square (indicative of a reward) or a red square and exploded balloon (indicative of loss) appeared after the pumps accompanied by an auditory feedback played 500ms after the visual feedback. Visual feedback lasted 1000ms followed by a 1000-1200ms crosshair and a 100ms blank screen before the next balloon was presented. The total points earned, balloon/trial number, and the explosion point for the last balloon were displayed at the bottom of the screen. After the feedback, a new uninflated balloon appeared on screen until a total of 60 balloons were completed.
Change of Objective Cognitive Performance (Delay Discounting Task) | Baseline, one week after the intervention and 6-month after the intervention
  In the delay discounting task, participants are asked to choose between two options: an immediate smaller reward (e.g., $17 now) and a later larger reward (e.g., $20 in 5 months). The magnitude of the immediate smaller reward and the magnitude and delay of the later larger reward varies from trial to trial. The immediate smaller option is always smaller and earlier than the later larger option. Performance indicator: The area under the curve (AUC) method will be used to analyse the data. A smaller AUC value indicates a higher impulsive choice.
Change of Objective Cognitive Performance (Information Sampling Task) | Baseline, one week after the intervention and 6-month after the intervention
  In the information sampling task, participants are presented with a matrix of 25 gray boxes and 2 larger colored panels (yellow and blue) at the bottom. When participants touch a gray box, it will open to show its color (yellow or blue). Participants are instructed to decide which color they think is in the majority. It is up to the participants how many boxes they would like to open before making the decision. There are two conditions, i.e., Fixed win condition and Decreasing Win condition, each consisting of 10 trials. Performance indicators: The mean probability of being correct at the point of decision (P correct), the mean number of boxes opened per trial, as well as discrimination and sampling errors will be analysed. The lower mean P correct reflects higher reflection impulsivity.
Change in ERP components on the Cued Go/NoGo task | Baseline, one week after the intervention and 6-month after the intervention
  The ERP components including CNV, NoGo N2, and NoGo P3 will be examined between the treatment group and control, in baseline, post-treatment and followup sessions.
Change in ERP components on the Balloon Analogue Risk Task | Baseline, one week after the intervention and 6-month after the intervention
  The ERP components including feedback-related negativity (FRN) and P300 amplitudes to both negative and positive feedback will be examined on the Balloon Analogue Risk Task.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Clinic and Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong